CLINICAL TRIAL: NCT04972773
Title: Spinal Cord Injury Mental Health Functional Outcomes Improved by Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Karen Smith, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RMED-087-21
Record Dates: First submitted 2021-06-30; First posted 2021-07-22 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries; Mindfulness Meditation; Mental Health Wellness 1
Keywords: Spinal Cord Injuries; Mindfulness meditation; Mental Health outcomes; Quality of life
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Treatment: Computer-based randomization (https://www.randomizer.org/) will assign half of the participants taken in on a rolling basis to a MM intervention group (in addition to standard-therapy) and half of the participants to the standard-therapy control group which run in parallel.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will be established by having a separate collaborator randomize participants to one of the two arms and manage the notification of participants of their allocation, while the primary investigator and outcomes assessor is not informed of this randomization.
  Only the researchers will be blinded to a subject's group. Because of the nature of asking the intervention group, but not the control group, to complete additional MM practice, the participants will not be blinded. Thus no provisions need to be made to break the code of the blinding protocol in an emergency. The researchers (investigator and outcomes assessors) will be unaware of participants group assignment, so as not to show preference to one group. The master code that connects participant data to a participant ID will be stored separately from the rest of the data on a USB, otherwise keeping researchers blind to the participant's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MM + standard-therapy intervention group (Experimental): In addition to receiving standard-therapy, participants will be asked to practice MM using a MM app for at least 10 minutes per day from weeks 0 to 8.
  Interventions: Behavioral: Mindfulness meditation (MM)
- Standard-therapy control group (No Intervention): Participants randomized to the standard-therapy control group will receive their typical in- or out-patient therapy. This is expected to include small doses of MM.

INTERVENTIONS:
Behavioral: Mindfulness meditation (MM) — Towards this additional MM practice, participants will be able to use any combination of the MM apps: "Insight timer", which focuses on community/group-like therapy, "Healthy minds", which focuses on resilience that is essential in disability adjustment, and "Smiling mind", that reminds patients of their family/support structures. These three options were chosen for delivering free MM with different focuses that would cater to the variety of SCI patients needs. Participants will be alerted if they are not achieving 30 minutes of additional MM per week. This will guarantee that the treatment group have a higher time spent on MM for dose-response analysis. Participants will receive a reminder email (see attached) on the Sunday evening of a week with <30 minutes of additional MM encouraging them to use their mindfulness app.
  Other Names: Consumer app-based meditation; Insight timer; Healthy minds; Smiling mind
  Arms: MM + standard-therapy intervention group

SUMMARY:
Recovery from injury is an immune function but also involves stress. Spinal cord injury (SCI) patients are one population with a difficult recovery journey. Improvements in SCI rehabilitation could benefit patient's recovery and decrease their functional limitations. Lack of independence and chronic pain contributes to a higher rate of mental health problems (48.5%) and clinical stress (25%) in SCI patients. Depression is more common among auto-immune phenotypes and depression patients have higher pro-inflammatory cytokine profiles, suggesting stress impacts the immune system and thus opposes recovery. Mindfulness meditation (MM) is one form of stress-reduction therapy, which also decreases anxiety, depression, and pain. Little research has investigated whether this extends to functional outcomes of mental health during recovery. The investigators will look at the "functional outcomes of mental health", including stress, pain, quality of life, quality of sleep, and outcomes of depression using validated surveys. The investigators hypothesize that MM will significantly improve functional outcomes of mental health in SCI patients during their rehabilitation in a dose-dependent fashion, compared to 'standard therapy' alone control, with effects sustained 1-month post-intervention. Patients will take surveys of their mindfulness practices and mental health functional outcomes at 0 weeks (baseline), 8 weeks (post-treatment), and 12 weeks (follow-up). MM will be delivered to a randomized sample of SCI patients via one of three MM apps for 8 weeks. Linear regression will identify if patients practicing more MM have better mental health functional outcomes in a dose-dependent manner. The findings from this study will provide evidence of sustained stress-relief and mental health functional outcomes of consumer-based MM apps, which can be applied to improve SCI rehabilitation in an accessible manner.

DETAILED DESCRIPTION:
SCI can pose significant limitations on a patient, with paralyzed patients requiring assisted living for activities of daily living like eating, dressing, hygiene, bathing, toileting, transferring and walking, any improvement in rehabilitation is important. Lack of independence and chronic pain contributes to a higher rate of mental health problems (48.5%) and clinical stress (25%) in these patients. Stress-targeted therapies like MM are correlated to better QOL, mental health, and moderately to physical health in other therapeutic populations. It is essential to translate these MM results on the functional outcomes of mental health to SCI patients. Effective early rehabilitation is essential to minimize muscle, bone, and flexibility loss and better stress management and pain control are key to getting into early rehabilitation. The stress and pain control MM could offer would benefit not only recovery but also health. New methods for pain management are essential because most current pain drugs are or become ineffective in up to half of patients or have strong side effects and/or societal burdens like opioids. Effective non-medication management of pain like MM could reduce opioid prescriptions and lessen the strain of addiction on society. This study aims not only to address the efficacy of MM on traditional outcome measures but also to examine the effect on functional outcomes, making it more clinically applicable.

In balancing limited resources like healthcare expenditure and healthcare professionals' time, MM mobile applications are one solution that promises accessible, cost-effective, and time-effective treatments, giving patients' autonomy and flexibility to incorporate mindfulness into their rehabilitation. MM present a promising, novel advancement to rehabilitation, stress control, and functional outcomes of mental health, that needs more research to apply in SCI patient groups through mobile app modalities.

Patients:

A participant will be eligible if they are an English-speaking adult in- or out-patient of all diagnoses in the SCI Rehabilitation Program at Providence Care Hospital or with SCI Ontario and own a smartphone on which they are willing to download a MM app. Sample size calculation identifies that 112 total participants are required to give 80% statistical power at a two-sided alpha of 0.05 for significance based on previous stress reduction effect size in SCI patients (n=56, 2 groups, N=112). Participants will be enrolled for 12 weeks, 8 of which will be the treatment weeks and 4 of which will be the follow-up weeks.

Treatment:

Computer-based randomization (https://www.randomizer.org/) will assign half of the participants to a MM intervention group (in addition to 'standard therapy') and half of the participants to the 'standard therapy' control group. Randomization will be stratified by in-/out-patient as the in-patients receive some MM as a part of 'standard therapy', while the out-patients do not. The goal of randomization and adding MM as a treatment is to ensure a distribution of doses of MM for analysis. Analysis of the data for a dose-dependent response will combat inherent contamination in the control group as a small amount of MM is a part of standard therapy for in-patients.

'Standard therapy' control group: Participants randomized to the 'standard therapy' control group will receive their typical in- or out-patient therapy. This is expected to include small doses of MM.

Intervention group: Participants randomized to the intervention group, in addition to receiving 'standard therapy', will be asked to practice MM using a MM app for at least 10 minutes per day from weeks 0 to 8. Towards this additional MM practice, participants will be able to use any combination of the MM apps: "Insight timer", which focuses on community/group-like therapy, "Healthy minds", which focuses on resilience that is essential in disability adjustment, and "Smiling mind", that reminds patients of their family/support structures. These three options were chosen for delivering free MM with different focuses that would cater to the variety of SCI patients needs. Participants will be alerted if they are not achieving 30 minutes of additional MM per week. This will guarantee that the treatment group have a higher time spent on MM for dose-response analysis. Participants will receive a reminder email (see attached) on the Sunday evening of a week with <30 minutes of additional MM encouraging them to use their mindfulness app.

Measurements:

Demographic data (age, injury type, mental health history, medication use, and therapy/counselling history) and current and a 1-year history of mindfulness practices, including use of MM apps, yoga, group MM, CBT, and MM technique use like body scan will be collected at baseline (0 weeks).

Both groups (intervention and control) will receive a survey each week asking them to report their MM practice total time for the week as a way of monitoring their MM dose.

Additionally, both groups will be assessed using Qualtrics at baseline, post-intervention (8 weeks), and at follow-up (12 weeks) for the outcome measures of:

* Mindfulness via the 39-item Five Facet Mindfulness Questionnaire (FFMQ)
* Anxiety and depression via the 14-item Hospital Anxiety and Depression Scale (HADS), validated in SCI
* Functional outcomes of mental health, including:

  * Stress via the 10-item Perceived Stress Scale survey
  * Quality of life (QOL) via the 26-item WHO QOL-BREF measuring physical health, psychological health, social relationships, and health of the patient's environment, validated in SCI
  * Quality of Sleep via the Pittsburgh Sleep Quality Index (PSQI)
  * Pain via the Global Pain Scale and its outcomes via the validated 13-item Pain catastrophizing scale
  * Depression outcomes via the validated Clinical Global Impression - Clinical Improvement tool, as recommended for quantifying the mental health outcomes Finally, in only the intervention group, feasibility will be measured via adherence (in minutes/week) to the prescribed 10 min/day of MM for 8 weeks and acceptability will be measured via a Likert-scale (1-5) satisfaction survey delivered in week 8.

Statistical analysis:

All statistical analyses will be performed in GraphPad Prism 7 (GraphPad Software Inc., CA, USA). First, all data will be examined for distribution normality and outliers to ensure that statistical tests hold validity.

Group data (n=56) will be normalized to baseline and then averaged for comparison. The analysis will compare the Likert scale-based outcomes of mindfulness, anxiety and depression, stress, QOL, quality of sleep, pain, and depression outcomes between the intervention (high dose) and control (low dose) group at the three time points (2x3 analysis). Statistical significance will be tested using a two-way sample t-test in all experiments, where a P-value of =0.05 will be considered statistically significant between groups. The Bonferroni method to correct for multiple comparisons with a Bonferonni a=0.016 for within-group comparison will be used. The Cohen d effect size will be reported. To analyze the dose-dependent effects of MM, MM time will be treated as a continuous variable. General linear models can be used to compare functional outcomes of mental health based on MM dose at the post-intervention (8 week) measurement. A linear mixed-model will test the sustained mean difference between groups and time with group×time as an interaction factor at follow-up (12 week).

Feasibility will be assessed by calculating adherence to the treatment protocol as a percentage of participants and as a percentage of individual's time spent doing MM based on weekly self-reports by participants of their MM activities. Acceptability will be calculated by averaging responses to the satisfaction survey (rating 1-5) for those assigned to the MM intervention group.

Data presentation:

Data will be graphed as mean±sem of each outcome measure vs time engaged with MM, with the control group naturally being at a deficit to the intervention group to illustrate any dose-dependent effects of MM.

The primary aims of this research are:

1) Beyond the negative effect of stress on mental health, mental health negatively affects physical health via poor sleep, less exercise, and unhealthy eating. Yet, little research exists on mental health functional outcomes and it remains controversial. Despite the importance of QOL, metanalysis found this was not an outcome in most studies and only 5% of studies look at functional outcomes of mental health. This research aims to measure functional outcomes of mental health by measuring QOL, stress, pain, depression/anxiety, and depression disability.

The secondary aims of this research are:

1. Most studies use heterogenous injury type and severity, preventing meaningful statistical comparison. While evidence exists for CLBP, no evidence yet exists for MM effects in SCI. This research will isolate SCI patients to understand the effects of MM.
2. Research focuses on programs like mindfulness-based stress reduction (MBSR), an 8-week group MM program. Although effective, these formalized programs are less feasible during social distancing, cost more time and money, and cannot serve outpatients. This research will focus on a modality of MM that is convenient, cost-effective, and accessible, but has precedent in the literature - mobile MM apps, including "Insight timer", "Healthy minds", and "Smiling mind". Mobile health apps offer remote care, user autonomy, and longer treatment. However, these apps require independent testing for efficacy and feasibility. This study hopes to make MM more accessible by assessing the outcomes of MM app use.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* legal adults (age > 17)
* in- or out-patients of all diagnoses in the SCI Rehabilitation Program at Providence Care Hospital or with SCI Ontario (ie. have SCI)
* own a smartphone on which they are willing to download the MM app(/s)
* have hand function or can provide a caregiver themselves to assist them with filling out 1 hour of questionnaires at three different time points in the study (0 weeks, 8 weeks, and 12 weeks)
* ability to consent themselves to research

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Change in Mindfulness during treatment phase assessed via the 39-item Five Facet Mindfulness Questionnaire (FFMQ) | Weeks 0-8 (treatment [or control])
  With 5 categories: 1) Observe, 2) Describe, 3) Act with Awareness, 4) Non-judge, each of which is on a scale of 8-40 where greater is more mindful and 5) Non-react, which is on a scale of 7-35 where greater is more mindful
Change in Anxiety and depression during treatment phase assessed via the 14-item Hospital Anxiety and Depression Scale (HADS) | Weeks 0-8 (treatment [or control])
  With two categories: 1) Depression, 2) Anxiety, each of which can range from 0-21, where an increased score is more deviation from neurotypical (depressed or anxious)
Change in Stress during treatment phase assessed via the 10-item Perceived Stress Scale survey | Weeks 0-8 (treatment [or control])
  With a range of 0-40 with higher scores being more stress
Change in Quality of life during treatment phase assessed via the 26-item World Health Organization (WHO) Quality of life (QOL)-Abbreviated (BREF) | Weeks 0-8 (treatment [or control])
  Measuring physical health, psychological health, social relationships, and health of the patient's environment, validated in SCI patients, averaged responses (as oppose to summed) ranging from 1 - 5, where 5 is a higher quality of life
Change in Quality of Sleep during treatment phase assessed via the Pittsburgh Sleep Quality Index (PSQI) | Weeks 0-8 (treatment [or control])
  With a range of 0-21 points, where higher scores indicate more sleep disturbances
Change in Pain during treatment phase assessed via the validated Global Pain Scale | Weeks 0-8 (treatment [or control])
  With a range of 0-100, where 100 is greater global (physical, emotional, functional, and clinical) pain
Change in Pain Catastrophizing during treatment phase assessed via the validated 13-item Pain catastrophizing scale | Weeks 0-8 (treatment [or control])
  With a range of 0 - 52, where higher values indicate more catastrophizing about pain
Change in Clinical Improvement of Depression during treatment phase assessed via the validated Clinical Global Impression - Clinical Improvement tool | Weeks 0-8 (treatment [or control])
  Which has items: 1) Severity of illness, range 1 - 7, with greater being more severe. 2) Global improvement, range 1 - 7, with greater being more worsening and lesser being more improvement. 3) Efficacy, range 0.25 - 4 based on the multiplication of the two answers - for therapeutic effect, the response: "Marked improvement" = 2, "Moderate improvement" = 1.5, "Minimal improvement" = 1, or "Worse" = 0.5; the while response: "No side effects" multiples the result by 2, "Side effects which don't interfere with functioning" multiplies the result by 1, "Side effects which significantly interfere with patient's functioning" multiples the result by 0.66X, and "side effects worse than the benefits" multiples the result by 0.5. Lower scores indicate worse clinical outcome (no effect or too many side effects), higher scores mean better outcome (effects and few side effects), with 1 being the cut-off for clinical recommendation
Change in Mindfulness during follow-up phase assessed via the 39-item Five Facet Mindfulness Questionnaire (FFMQ) | Weeks 8-12 (follow-up)
  With 5 categories: 1) Observe, 2) Describe, 3) Act with Awareness, 4) Non-judge, each of which is on a scale of 8-40 where greater is more mindful and 5) Non-react, which is on a scale of 7-35 where greater is more mindful
Change in Anxiety and depression during follow-up phase assessed via the 14-item Hospital Anxiety and Depression Scale (HADS) | Weeks 8-12 (follow-up)
  With two categories: 1) Depression, 2) Anxiety, each of which can range from 0-21, where an increased score is more deviation from neurotypical (depressed or anxious)
Change in Stress during follow-up phase assessed via the 10-item Perceived Stress Scale survey | Weeks 8-12 (follow-up)
  With a range of 0-40 with higher scores being more stress
Change in Quality of life during follow-up phase assessed via the 26-item World Health Organization (WHO) Quality of life (QOL)-Abbreviated (BREF) | Weeks 8-12 (follow-up)
  Measuring physical health, psychological health, social relationships, and health of the patient's environment, validated in SCI patients, averaged responses (as oppose to summed) ranging from 1 - 5, where 5 is a higher quality of life
Change in Quality of Sleep during follow-up phase assessed via the Pittsburgh Sleep Quality Index (PSQI) | Weeks 8-12 (follow-up)
  With a range of 0-21 points, where higher scores indicate more sleep disturbances
Change in Pain during follow-up phase assessed via the validated Global Pain Scale | Weeks 8-12 (follow-up)
  With a range of 0-100, where 100 is greater global (physical, emotional, functional, and clinical) pain
Change in Pain Catastrophizing during follow-up phase assessed via the validated 13-item Pain catastrophizing scale | Weeks 8-12 (follow-up)
  With a range of 0 - 52, where higher values indicate more catastrophizing about pain
Change in Clinical Improvement of Depression during follow-up phase assessed via the validated Clinical Global Impression - Clinical Improvement tool | Weeks 8-12 (follow-up)
  Which has items: 1) Severity of illness, range 1 - 7, with greater being more severe. 2) Global improvement, range 1 - 7, with greater being more worsening and lesser being more improvement. 3) Efficacy, range 0.25 - 4 based on the multiplication of the two answers - for therapeutic effect, the response: "Marked improvement" = 2, "Moderate improvement" = 1.5, "Minimal improvement" = 1, or "Worse" = 0.5; the while response: "No side effects" multiples the result by 2, "Side effects which don't interfere with functioning" multiplies the result by 1, "Side effects which significantly interfere with patient's functioning" multiples the result by 0.66X, and "side effects worse than the benefits" multiples the result by 0.5. Lower scores indicate worse clinical outcome (no effect or too many side effects), higher scores mean better outcome (effects and few side effects), with 1 being the cut-off for clinical recommendation

SECONDARY OUTCOMES:
Average Adherence as a marker of how feasibly a patient can complete the mindfulness dose requested by the protocol | Weekly for 8 weeks
  Measuring adherence (in minutes/week) as = actual time doing mindfulness / the prescribed total (70 mins/week, since 10 min/day of MM), reported as a percentage which can range from 0%-above 100%, where higher values indicate greater adherence and thus suggest greater feasibility. Results will be averaged over the 8 weeks.
Self-reported Likert-scale rating of satisfaction with the mindfulness meditation practice as a measure of acceptability | Week 8
  Assessed via a Likert-scale ranging from 1-5 on a satisfaction survey, where a higher value indicates greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith, MD, Principal Investigator — Queen's University
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Migliorini C, Tonge B, Taleporos G. Spinal cord injury and mental health. Aust N Z J Psychiatry. 2008 Apr;42(4):309-14. doi: 10.1080/00048670801886080. PMID 18330773
- [Background] Maldonado Bouchard S, Hook MA. Psychological stress as a modulator of functional recovery following spinal cord injury. Front Neurol. 2014 Apr 9;5:44. doi: 10.3389/fneur.2014.00044. eCollection 2014. PMID 24782818
- [Background] Tran J, Dorstyn DS, Burke AL. Psychosocial aspects of spinal cord injury pain: a meta-analysis. Spinal Cord. 2016 Sep;54(9):640-8. doi: 10.1038/sc.2016.66. Epub 2016 May 10. PMID 27163453
- [Background] Pillastrini P, Mugnai R, Bonfiglioli R, Curti S, Mattioli S, Maioli MG, Bazzocchi G, Menarini M, Vannini R, Violante FS. Evaluation of an occupational therapy program for patients with spinal cord injury. Spinal Cord. 2008 Jan;46(1):78-81. doi: 10.1038/sj.sc.3102072. Epub 2007 Apr 24. PMID 17453011
- [Background] Krupa T, Fossey E, Anthony WA, Brown C, Pitts DB. Doing daily life: how occupational therapy can inform psychiatric rehabilitation practice. Psychiatr Rehabil J. 2009 Winter;32(3):155-61. doi: 10.2975/32.3.2009.155.161. PMID 19136347
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Hearn JH, Cross A. Mindfulness for pain, depression, anxiety, and quality of life in people with spinal cord injury: a systematic review. BMC Neurol. 2020 Jan 21;20(1):32. doi: 10.1186/s12883-020-1619-5. PMID 31964353
- [Background] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Background] Hearn JH, Finlay KA. Internet-delivered mindfulness for people with depression and chronic pain following spinal cord injury: a randomized, controlled feasibility trial. Spinal Cord. 2018 Aug;56(8):750-761. doi: 10.1038/s41393-018-0090-2. Epub 2018 Mar 26. PMID 29581519